CLINICAL TRIAL: NCT00848198
Title: A Prospective Study to Establish Normative Values, Demographic Variations, Referent Diagnostic Values and Disease Severity Correlations for Dry Eye Disease and TearLab Osmometry.
Brief Title: TearLab Core Validation Study to Establish Referent Values for Dry Eye Disease
Acronym: CVS
Status: Completed | Type: Observational
Sponsor: TearLab Corporation (Industry)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: TP00007 OTO
Record Dates: First submitted 2009-02-18; First posted 2009-02-20 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: Dry Eye Disease; Dry Eye Syndrome; Dry Eye
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal: Subjects with no objective signs of Dry Eye Disease
- Dry Eye Disease: Subjects with objective signs of Dry Eye Disease

SUMMARY:
This is a prospective, observational case series to determine the clinical utility of tear osmolarity and other commonly used objective tests to diagnose dry eye disease, as well as to establish referent values for objective tests of the disease.

DETAILED DESCRIPTION:
This is a prospective, observational case series to determine the clinical utility of tear osmolarity, tear film breakup time, corneal fluorescein staining, conjunctival lissamine green staining, Schirmer's test without anesthesia, Bron/Foulks meibomian glan grading and the ocular surface disease index to diagnose dry eye disease, as well as to establish referent values for objective tests of the disease. Patients were recruited across sites in the EU and US from the general clinical population.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 79 years of age.
* Must understand and be able, willing and likely to fully comply with study procedures and restrictions.

Exclusion Criteria:

* Clinically significant eyelid deformity or eyelid movement disorder that is caused by conditions such as notch deformity, incomplete lid closure, entropion, ectropion, hordeola or chalazia..
* Previous ocular disease leaving sequelae or requiring current topical eye therapy other than for Dry Eye Disease, including, but not limited to: active corneal or conjunctival infection of the eye and ocular surface scarring.
* Active ocular allergy.
* LASIK or PRK surgery that was performed within one year of Visit 1.
* Started or changed the dose of chronic ocular medication within 30 days of visit 1.
* Contact lens worn within the past eight (8) hours.
* Any ophthalmologic drops within 2 hours of screening and visit 1 procedures.
* Pregnancy or lactation.
* Abnormality of nasolacrimal drainage (by history).
* Punctual plugs placement or cauterization within 30 days of Visit 1
* Started or changed the dose of chronic systemic medication known to affect tear production including, but not limited to antihistamines, antidepressants, diuretics, corticosteroids or immunomodulators within 30 days of Visit 1.
* Systemic disease known to affect tear production or loss including, but not limited to thyroid eye disease, that has been diagnosed or has not been stable within 30 days of Visit 1.
* Known hypersensitivity to any of the agents used in testing i.e. sodium fluorescein, lissamine green, oxybuprocaine or proparacaine.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmology and Optometry Clinics
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Foulks, MD, Study Chair — Kentucky Lions Eye Center, University of Louisville
Locations (10):
- United States (6):
  - Gordon Binder Weiss Vision Institute, San Diego, California
  - Kentucky Lion Eye Center, Louisville, Kentucky
  - Pepose Vision Institute, Chesterfield, Missouri
  - Tauber Eye Clinic, Kansas City, Missouri
  - Mundorf Eye Center, Charlotte, North Carolina
  - Ohio State University, Columbus, Ohio
- Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris, France
- University of Wurzburg, Würzburg, Germany
- Hospital Clinico San Carlos, Madrid, Spain
- Division of Vision Sciences, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data was published in AJO May 2011 and IOVS Dec.2010.

REFERENCES:
- [Result] Lemp MA, Bron AJ, Baudouin C, Benitez Del Castillo JM, Geffen D, Tauber J, Foulks GN, Pepose JS, Sullivan BD. Tear osmolarity in the diagnosis and management of dry eye disease. Am J Ophthalmol. 2011 May;151(5):792-798.e1. doi: 10.1016/j.ajo.2010.10.032. Epub 2011 Feb 18. PMID 21310379
- [Result] Sullivan BD, Whitmer D, Nichols KK, Tomlinson A, Foulks GN, Geerling G, Pepose JS, Kosheleff V, Porreco A, Lemp MA. An objective approach to dry eye disease severity. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6125-30. doi: 10.1167/iovs.10-5390. Epub 2010 Jul 14. PMID 20631232
- [Derived] Lemp MA, Crews LA, Bron AJ, Foulks GN, Sullivan BD. Distribution of aqueous-deficient and evaporative dry eye in a clinic-based patient cohort: a retrospective study. Cornea. 2012 May;31(5):472-8. doi: 10.1097/ICO.0b013e318225415a. PMID 22378109

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects between the ages of 18 and 82 years were included in the study. Participants were chosen from 10 sites in the E.U. and U.S. from the general patient population. 314 total subjects were enrolled.
Pre-assignment Details: Of the first 314 subjects enrolled, only 299 (n = 218 female, n = 81 male), were used in the analysis with the remainder disqualified for incomplete case report forms and lack of data from the single visit.
Groups:
- Total Number of Participants: All participants who were tested using common signs and symptoms for dry eye disease
Period: Overall Study
Arm/Group | Total Number of Participants
Started | 314
Completed | 299
Not Completed | 15
Not completed — Incomplete Case Report Forms | 15

BASELINE CHARACTERISTICS:
Arm/Group | Total Number of Participants
Number analyzed (Participants) | 314
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 269
  >=65 years | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233
  Male | 81
Region of Enrollment [Number; unit: participants]
  France | 50
  United States | 139
  Spain | 50
  Germany | 50
  United Kingdom | 25

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Test Data for Disease Using Tear Osmolarity Threshold > 308 mOsm/L
Description: Tear osmolarity was measured with a laboratory-on-a-chip, to simultaneously collect and analyze the electrical impedance of a 50 nL tear sample from the interior lateral meniscus (TearLab Osmolarity System). A cutoff threshold of more than 308 mOsm/L was used for differentiating normal from mild to moderate subjects.
  The clinical tools most commonly used in grading dry eye severity are symptomatology (e.g. questionnaires such as the Ocular Surface Disease Index (OSDI) or McMonnies Dry Eye Questionnaire), tear osmolarity, tear film breakup time (TBUT), fluoresceine or lissamine green staining of the cornea and conjunctiva, meibomiam secretion scoring, and the Schirmer test.To convert all the various clinical measurements into a common unit system, based on their breakpoints provided by the Dry Eye Workshop (DEWS), a composite score was created. Its scale being between 0 (representing the least evidence of disease) and 1 (representing the most evidence of disease).
Time Frame: Single visit
Measure: Number; unit: participants
Groups:
- Participants With Dry Eye Disease: Presence of dry eye disease as defined by positive reference test
- Participants Without Dry Eye Disease (Normal): Absence of dry eye disease as defined by negative reference test
Arm/Group | Participants With Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 224 | 75
participants
  Positive diagnostic test | 177 | 14
  Negative diagnostic test | 47 | 61
Statistical Analysis 1: Comparison: Participants With Dry Eye Disease; Test type: Superiority or Other; Sensitivity = 87.1, 95% CI 2-sided [83.2 to 90.9]
Statistical Analysis 2: Comparison: Participants Without Dry Eye Disease (Normal); Test type: Superiority or Other; Specificity = 72.0, 95% CI 2-sided [66.9 to 77.1]

2. Primary Outcome: Diagnostic Test Data for Disease Using Schirmer Test Threshold < 7 mm
Description: A 5-minute Schirmer test was performed with sterile strips without anesthetic (Tear Flo). The cutoff threshold of <7mm was used to differentiating normal from mild subjects.
  The clinical tools most commonly used in grading dry eye severity are symptomatology (e.g. questionnaires such as the Ocular Surface Disease Index (OSDI) or McMonnies Dry Eye Questionnaire), tear osmolarity, tear film breakup time (TBUT), fluoresceine or lissamine green staining of the cornea and conjunctiva, meibomiam secretion scoring, and the Schirmer test. To convert all the various clinical measurements into a common unit system, based on their breakpoints provided by the Dry Eye Workshop (DEWS), a composite score was created. Its scale being between 0 (representing the least evidence of disease) and 1 (representing the most evidence of disease).
Time Frame: Single visit
Measure: Number; unit: participants
Arm/Group | Participants With Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 224 | 75
participants
  Positive diagnostic test | 89 | 13
  Negative diagnostic test | 135 | 62
Statistical Analysis 1: Comparison: Participants With Dry Eye Disease; Test type: Superiority or Other; Sensitivity = 39.7, 95% CI 2-sided [34.2 to 45.3]
Statistical Analysis 2: Comparison: Participants Without Dry Eye Disease (Normal); Test type: Superiority or Other; Specificity = 82.7, 95% CI 2-sided [78.4 to 87.0]

3. Primary Outcome: Diagnostic Test Data for Disease Using Tear Film Breakup Time Threshold < 5 Seconds
Description: Tear film breakup time was measured by instilling 5μL of a 2% sodium fluoresceine solution and calculating the average of three consecutive breakup times, manually determined with a stopwatch. The cutoff of <5 seconds was used to differentiate normal from dry eye subjects. The clinical tools most commonly used in grading dry eye severity are symptomatology (e.g. questionnaires such as the Ocular Surface Disease Index (OSDI) or McMonnies Dry Eye Questionnaire), tear osmolarity, tear film breakup time (TBUT), fluoresceine or lissamine green staining of the cornea and conjunctiva, Meibomiann secretion scoring, and the Schirmer test. To convert all the various clinical measurements into a common unit system, based on their breakpoints provided by the Dry Eye Workshop (DEWS), a composite score was created. Its scale being between 0 (representing the least evidence of disease) and 1 (representing the most evidence of disease).
Time Frame: Single visit
Measure: Number; unit: participants
Arm/Group | Participants With Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 224 | 75
participants
  Positive diagnostic test | 161 | 13
  Negative diagnostic test | 63 | 62
Statistical Analysis 1: Comparison: Participants With Dry Eye Disease; Test type: Superiority or Other; Sensitivity = 71.9, 95% CI 2-sided [66.8 to 77.0]
Statistical Analysis 2: Comparison: Participants Without Dry Eye Disease (Normal); Test type: Superiority or Other; Specificity = 82.7, 95% CI 2-sided [78.4 to 87.0]

4. Primary Outcome: Diagnostic Test Data for Disease Using Corneal Staining Threshold > Grade 4/15
Description: Corneal Staining was evaluated under cobalt blue illumination 2.5 to 3.0 minutes after fluorescein instillation. Staining amplitude followed the National Eye Institute/Industry Workshop scale. The cutoff threshold >4/15 was used to differentiate normals from dry eye subjects. The clinical tools most commonly used in grading dry eye severity are symptomatology (e.g. questionnaires such as the Ocular Surface Disease Index (OSDI) or McMonnies Dry Eye Questionnaire), tear osmolarity, tear film breakup time (TBUT), fluoresceine or lissamine green staining of the cornea and conjunctiva, meibomiam secretion scoring, and the Schirmer test.To convert all the various clinical measurements into a common unit system, based on their breakpoints provided by the Dry Eye Workshop (DEWS), a composite score was created. Its scale being between 0 (representing the least evidence of disease) and 1 (representing the most evidence of disease).
Time Frame: Single visit
Measure: Number; unit: participants
Arm/Group | Participants With Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 224 | 75
participants
  Positive diagnostic test | 61 | 1
  Negative diagnostic test | 163 | 74
Statistical Analysis 1: Comparison: Participants With Dry Eye Disease; Test type: Superiority or Other; Sensitivity = 27.2, 95% CI 2-sided [22.2 to 32.3]
Statistical Analysis 2: Comparison: Participants Without Dry Eye Disease (Normal); Test type: Superiority or Other; Specificity = 98.7, 95% CI 2-sided [97.4 to 100.0]

5. Primary Outcome: Diagnostic Test Data for Disease Using Conjunctival Staining Threshold > Grade 3/12
Description: Conjunctival staining was performed 2.5 to 3.0 minutes after instillation of 10 μL of a 1% sodium lissamine green dye. Conjunctival staining followed the National Eye Institute/Industry Workshop scale. A cutoff threshold of grade >3/12 was used to differentiate normal from dry eye subjects. The clinical tools most commonly used in grading dry eye severity are symptomatology (e.g. questionnaires such as the Ocular Surface Disease Index (OSDI) or McMonnies Dry Eye Questionnaire), tear osmolarity, tear film breakup time (TBUT), fluoresceine or lissamine green staining of the cornea and conjunctiva, meibomiam secretion scoring, and the Schirmer test. To convert all the various clinical measurements into a common unit system, based on their breakpoints provided by the Dry Eye Workshop (DEWS), a composite score was created. Its scale being between 0 (representing the least evidence of disease) and 1 (representing the most evidence of disease).
Time Frame: Single visit
Measure: Number; unit: participants
Arm/Group | Participants With Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 224 | 75
participants
  Positive diagnostic test | 115 | 4
  Negative diagnostic test | 109 | 71
Statistical Analysis 1: Comparison: Participants With Dry Eye Disease; Test type: Superiority or Other; Sensitivity = 51.3, 95% CI 2-sided [45.7 to 57.0]
Statistical Analysis 2: Comparison: Participants Without Dry Eye Disease (Normal); Test type: Superiority or Other; Specificity = 94.7, 95% CI 2-sided [92.1 to 97.2]

6. Primary Outcome: Diagnostic Test Data for Disease Using Meibomian Gland Grading Threshold > Grade 5/27
Description: Meibomian dysfunction was assessed to grade the quality, expressibility, and volume of gland secretion, according to Bron/Foulks scoring system. A cutoff threshold of grade 5/27 was used to differentiate normal from dry eye subjects. The clinical tools most commonly used in grading dry eye severity are symptomatology (e.g. questionnaires such as the Ocular Surface Disease Index (OSDI) or McMonnies Dry Eye Questionnaire), tear osmolarity, tear film breakup time (TBUT), fluoresceine or lissamine green staining of the cornea and conjunctiva, meibomiam secretion scoring, and the Schirmer test.To convert all the various clinical measurements into a common unit system, based on their breakpoints provided by the Dry Eye Workshop (DEWS), a composite score was created. Its scale being between 0 (representing the least evidence of disease) and 1 (representing the most evidence of disease).
Time Frame: Single visit
Measure: Number; unit: participants
Arm/Group | Participants With Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 224 | 75
participants
  Positive diagnostic test | 137 | 16
  Negative diagnostic test | 87 | 59
Statistical Analysis 1: Comparison: Participants With Dry Eye Disease; Test type: Superiority or Other; Sensitivity = 61.2, 95% CI 2-sided [55.6 to 66.7]
Statistical Analysis 2: Comparison: Participants Without Dry Eye Disease (Normal); Test type: Superiority or Other; Specificity = 78.7, 95% CI 2-sided [74.0 to 83.3]

7. Primary Outcome: Diagnostic Test Data for Disease Using Ocular Surface Disease Index Threshold > 15/100
Description: Ocular Surface Disease Index (OSDI) Questionnaire was used for symptoms assessment. A cutoff of 15/100 score was used to differentiate between normal and dry eye subjects. The clinical tools most commonly used in grading dry eye severity are symptomatology (e.g. questionnaires such as the Ocular Surface Disease Index (OSDI) or McMonnies Dry Eye Questionnaire), tear osmolarity, tear film breakup time (TBUT), fluoresceine or lissamine green staining of the cornea and conjunctiva, meibomiam secretion scoring, and the Schirmer test.To convert all the various clinical measurements into a common unit system, based on their breakpoints provided by the Dry Eye Workshop (DEWS), a composite score was created. Its scale being between 0 (representing the least evidence of disease) and 1 (representing the most evidence of disease).
Time Frame: Single visit
Measure: Number; unit: participants
Arm/Group | Participants With Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 224 | 75
participants
  Positive diagnostic test | 131 | 20
  Negative diagnostic test | 93 | 55
Statistical Analysis 1: Comparison: Participants With Dry Eye Disease; Test type: Superiority or Other; Sensitivity = 58.5, 95% CI 2-sided [52.9 to 64.1]
Statistical Analysis 2: Comparison: Participants Without Dry Eye Disease (Normal); Test type: Superiority or Other; Specificity = 73.3, 95% CI 2-sided [68.3 to 78.3]

8. Secondary Outcome: Referent Values for Tear Osmolarity
Time Frame: Single visit
Measure: Mean (Standard Deviation); unit: mOsm/L
Groups:
- Participants With Severe Dry Eye Disease: Subjects with composite severity score less than 0.20
- Participants With Mild/Moderate Dry Eye Disease: Subjects with composite severity score between 0.20 and 0.35
- Participants Without Dry Eye Disease (Normal): Subjects with composite severity score greater than 0.35
Arm/Group | Participants With Severe Dry Eye Disease | Participants With Mild/Moderate Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 75 | 149 | 75
mOsm/L | 336.4 (22.3) | 315.0 (11.4) | 302.2 (8.3)

9. Secondary Outcome: Referent Values for Schirmer Test
Time Frame: Single visit
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Participants With Severe Dry Eye Disease | Participants With Mild/Moderate Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 75 | 149 | 75
mm | 8.2 (8.4) | 13.9 (9.5) | 19.3 (10.4)

10. Secondary Outcome: Referent Values for Tear Film Breakup Time
Time Frame: Single visit
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Participants With Severe Dry Eye Disease | Participants With Mild/Moderate Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 75 | 149 | 75
seconds | 2.7 (1.5) | 6.1 (4.9) | 11.8 (6.4)

11. Secondary Outcome: Referent Values for Corneal Staining
Description: Corneal Staining is used to identify and evaluate ocular surface and corneal damages. It was evaluated under cobalt blue illumination 2.5 to 3.0 minutes after fluorescein instillation. Staining amplitude followed the National Eye Institute/Industry Workshop scale. The cutoff threshold >4/15 was used to differentiate normals from dry eye subjects. A score of 0 indicates no damage of ocular surface/cornea, while the maximum for the most severe damage is 15.
Time Frame: Single visit
Measure: Mean (Standard Deviation); unit: Grade
Arm/Group | Participants With Severe Dry Eye Disease | Participants With Mild/Moderate Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 75 | 149 | 75
Grade | 5.1 (4.1) | 1.7 (1.9) | 0.4 (0.9)

12. Secondary Outcome: Referent Values for Conjunctival Staining
Description: Conjunctival staining is used to identify and evaluate dead or injured conjunctival cells. Conjunctival staining was performed 2.5 to 3.0 minutes after instillation of 10 μL of a 1% sodium lissamine green dye. Conjunctival staining followed the National Eye Institute/Industry Workshop scale. A cutoff threshold of grade >3/12 was used to differentiate normal from dry eye subjects. A score of 0 indicates no damage of conjunctival cells, while the maximum for the most severe damage is 12.
Time Frame: Single visit
Measure: Mean (Standard Deviation); unit: Grade
Arm/Group | Participants With Severe Dry Eye Disease | Participants With Mild/Moderate Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 75 | 149 | 75
Grade | 5.9 (3.6) | 2.6 (1.9) | 1.1 (1.4)

13. Secondary Outcome: Referent Values for Meibomian Gland Grading
Description: Meibomian gland dysfunction was assessed to grade the quality, expressibility, and volume of gland secretion, according to Bron/Foulks scoring system. A score of 0 indicates full integrity of these glands while the maximum of 27, is used for severe damage.
Time Frame: Single visit
Measure: Mean (Standard Deviation); unit: Grade
Arm/Group | Participants With Severe Dry Eye Disease | Participants With Mild/Moderate Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 75 | 149 | 75
Grade | 10.4 (5.2) | 5.6 (4.7) | 2.6 (2.7)

14. Secondary Outcome: Referent Values for Ocular Surface Disease Index
Description: Ocular Surface Disease Index (OSDI) Questionnaire was used for symptoms assessment and the index is calculated based on the responses given by the subject. A cutoff of 15/100 score was used to differentiate between normal and dry eye subjects. A score of 0 confirms no dry eye symptoms are present, while a maximum of 100 indicates the maximum severity of symptoms experienced by subjects.
Time Frame: Single visit
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Participants With Severe Dry Eye Disease | Participants With Mild/Moderate Dry Eye Disease | Participants Without Dry Eye Disease (Normal)
Number analyzed (Participants) | 75 | 149 | 75
Score | 41.2 (21.6) | 21.0 (19.2) | 5.5 (7.4)

ADVERSE EVENTS:
Time Frame: Time of the single visit
Description: No side effects were reported or observed.
Arm/Group | Total Number of Participants
Serious Adverse Events (participants affected / at risk) | 0/314
Other Adverse Events (participants affected / at risk) | 0/314

LIMITATIONS AND CAVEATS:
95/299 subjects were using topical medication at the time of measurement, potentially lowering the diagnostic performance of osmolarity (osmolarity is lowered and responds before the other tests during therapy) and compressing the referent spread.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No